CLINICAL TRIAL: NCT03067545
Title: Do Simple Running Technique Changes Reduce Pain and Change Injury Causing Mechanics in Runners With Common Running Related Injuries?
Brief Title: Do Simple Running Technique Changes Reduce Pain and Change Injury Causing Mechanics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salford (Other)
Responsible Party: Principal Investigator, Christopher Bramah, Principal Investigator, University of Salford
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSCR 16-49
Record Dates: First submitted 2017-02-17; First posted 2017-03-01 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Patellofemoral Pain Syndrome; Medial Tibial Stress Syndrome; Iliotibial Band Syndrome; Achilles Tendinopathy
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Medial Tibial Stress Syndrome; Iliotibial Band Syndrome

STUDY DESIGN:
Intervention Model Description: single subject repeated measures design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- step rate increase (Experimental): increase in running stride rate by 10%
  Interventions: Other: Step rate increase

INTERVENTIONS:
Other: Step rate increase — increase the step rate during running by 10% steps per minute

SUMMARY:
This project aims to investigate whether an increase in step rate can be used to reduce pain and injury causing movement patterns in runners who are currently experiencing achilles tendonopathy, iliotibial band syndrome, patellofemoral pain syndrome and medial tibial stress syndrome.

Many injuries have been reported to share similar injury causing movement patterns. For example iliotibial band syndrome and patellofemoral pain syndrome have been reported to be caused by increased side to side drop of the pelvis and inward movement of the hip.

Gait retraining is a method of changing the way people run in order to change movement patterns.Increasing step rate may present a gait retraining method that does not pose further injury risks and can be used across multiple different injury populations. Studies have shown increasing step rate can reduce frontal plane movement patterns at the pelvis, hip and foot as well as reducing sagittal plane joint angles such as ankle dorsiflexion. Based on the changes in movement patterns increasing step rate has been recommended as an intervention for the treatment of patellofemoral pain syndrome, medial tibial stress syndrome, iliotibial band syndrome and achilles tendonopathy. Therefore this study aims to investigate whether an increase in step rate can reduce pain and change injury causing mechanics in runners currently running with patellofemoral pain syndrome, iliotibial band syndrome, medial tibial stress syndrome or achilles tendinopathy.

The aim of the project is to use a simple gait intervention, increasing step rate to investigate if this technique change can reduce pain immediately, at short term follow up and long term follow up. The project will also look at whether an increased step rate can be maintained at follow up and whether this changes movement patterns proposed to be the cause of injury.

Runners will be recruited from local running clubs and competitions using poster advertisement at running clubs and emailed to running clubs

DETAILED DESCRIPTION:
All data will be collected at the university of Salford podiatry clinic gait laboratory. Participants will be recruited from running clubs and races via poster advertisement sent via email to the running club and on advertisement at the club. Also participants presenting at the running performance clinic with patellofemoral pain syndrome, iliotibial band syndrome, medial tibial stress syndrome and achilles tendonopathy will be invited to take part in the research study investigating the effects of gait retraining on injury. Participants who agree to take part will be sent an email confirming their appointment along with an information sheet detailing the study which they are encouraged to read before attending the appointment. They will have contact details of the lead researcher should they wish to ask any further questions

The objectives above will be addressed via the following data collection procedure:

On arriving at the running clinic participants will be informed that the gait retraining intervention aims to reduce pain when running and that there is a risk that the retraining protocol will not affect their pain. If there are no improvements to symptoms following gait retraining they will be then directed to the appropriate medical service for further management. Participants will be informed as to the procedures and given the chance to read through an information sheet again detailing the procedures involve. If on reading the information sheet participants do not wish to take part they can terminate the appointment at any time. Before data collection begins participants will sign a consent form, a running history form and a health screening questionnaire will be completed by a qualified physiotherapist in order to assess the patients suitability to complete the assessment with no further risk to their health.

Procedures:

Participants will attend two visits 4 weeks apart. The first visit will consist of an initial assessment data collection and a retraining session. Detailed below. The second visit will consist of the same procedures in the initial assessment.

Initial Assessment data collection:

Participants will complete the appropriate self reported outcome measure: if iliotibial band syndrome or patellofemoral pain syndrome they will complete the Lower extremity Functional Index and the Anterior Knee Pain Scale. If they present with medial tibial stress syndrome they will complete the medial tibial stress syndrome score and the Lower Extremity Functional Index. If they present with achilles tendonopathy they will complete the VISA - A score and the Lower Extremity Functional Index.

Before running retroreflective markers will be attached to the subject on specific points of their body: shoe, ankle joint, knee joint, greater trochanter of the hip, thigh, lower leg, pelvis (anterior superior iliac spine, posterior superior iliac spine, iliac crest), lumbar spine, thoracic spine, sternum and acromion process off the shoulders. This marker placement is according to a protocol previously established and validated in a project undertaken at the University of Salford. A qualysis motion capture system will then be used to track the movement of these markers as the participant runs on a treadmill. Once the marker data has been collected then we will use custom software to calculate the kinematic (joint movement) patterns for each person.

Participants are required to run on a treadmill at two different speeds (3.2, 3.8m/s). These speeds have been chosen based on running speeds used in previous research to allow comparability between studies. If participants feel they are unable to run at these speeds they can run at a self selected running speed.

They will be given a 6 minute accommodation period running on the treadmill at 3.2m/s. At this point data will then be collected for 1 minute of running in order to gain data for ten steps of running for the right and left feet. Speed will then be increased to 3.8m/s where they will be given a 1 minute accommodation period with data collected for a further minute of running.

A qualified physiotherapists will monitor the patients feels ok to continue at each 2 minute interval. At the end of data collection for each running speed the participant will be asked to rate their current level of pain on a scale of 0 = no pain to 10 = sever pain. If at any point the participants pain exceeds 8 out of 10 or the participant feels they can no longer continue running the data collection will be terminated.

Steps will be identified when the foot markers are in contact with the treadmill, once ten steps have been collected the data will be averaged across all trials for right and left feet. During the data collection injured participants will be asked to rate their current level of pain while running using a numerical rating scale 0 = no pain and 10 = sever pain.

Retraining Session:

Once data has been collected participants will then be asked to run for a further 5 minutes at each speed under an increased step rate condition with data collected for the final 1 minute of the trial. Step rate will be calculated as number of steps per minute. Step rate will then be increased by 10% and participants instructed to run to an audible metronome to ensure the step rate increase is achieved. Again at the end of each running speed participants will be asked to rate their current level of pain using a numerical rating scale.

Following data collection participants will be permitted up to a further 15 minute practise session running to maintain the increase in step rate without the metronome present to allow participants to adjust to the new running technique.

Participants will then be instructed to continue their current level of running using the new running technique. Participants will have contact details to the lead researcher (email and phone number) and will be requested to provide weekly updates regarding their running and if any pain is experienced. This will ensure patients are continuing to improve, not running with an increase in pain and are able to ask any questions they may have. If patient's symptoms are increasing they will be informed to stop running and terminated from the assessment and directed to the appropriate medical professional for further assessment.

Participants will be reassessed between 3 weeks and 5 weeks later following the same procedures outlined in the initial assessment data collection as well as at a 3 month follow up following the same procedures to investigate long term improvement.

ELIGIBILITY:
Inclusion Criteria:

* Runners presenting with patellofemoral pain syndrome, iliotibial band syndrome, medial tibial stress syndrome or achilles tendonopathy. Diagnosis to be confirmed via a qualified physiotherapist present at all sessions
* Currently running at self reported less than normal training volume
* Pain reported to onset during running
* Provide written consent to participate

Exclusion Criteria:

* history of a traumatic onset of injury
* previous lower limb surgery
* currently not running due to pain
* cardiac or respiratory disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
kinematic data (lower limb joint angles during running) | change from immediate, 4 weeks & 3 months
  lower limb joint angles during running
lower extremity functional scale | change from 4 weeks & 3 months
  patient reported outcome measure of lower limb pain symptoms
anterior knee pain scale | change from 4 weeks & 3 months
  patient reported outcome measure of lower limb pain symptoms
medial tibial stress syndrome score | change from 4 weeks & 3 months
  patient reported outcome measure of lower limb pain symptoms
numerical rating scale | change from 4 weeks & 3 months
  pain rating scale for pain experienced during running

SECONDARY OUTCOMES:
questionnaire measure of self reported running distance | change from 4 weeks & 3 months
  questionnaire measure of the total pain free distance the patient is able to run

CONTACTS AND LOCATIONS:
Overall Officials: Chris Bramah, MSc, Principal Investigator — University of Salford
Locations (1):
- University of Salford Health Sciences, Salford, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bramah C, Preece SJ, Gill N, Herrington L. A 10% Increase in Step Rate Improves Running Kinematics and Clinical Outcomes in Runners With Patellofemoral Pain at 4 Weeks and 3 Months. Am J Sports Med. 2019 Dec;47(14):3406-3413. doi: 10.1177/0363546519879693. Epub 2019 Oct 28. PMID 31657964